CLINICAL TRIAL: NCT00987805
Title: Efficacy of Banhasasim-tang on Functional Dyspepsia : a Randomized, Double Blind, Placebo Controlled, Two-center Trial
Brief Title: Efficacy of Banhasasim-tang on Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Jin-sung Kim, Full professor, Korea Health Industry Development Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B090029; ISRCTN51910678 (Other Grant/Funding Number: ISRCTN51910678)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Functional Dyspepsia
Keywords: Functional dyspepsia; Banhasasim-tang; Gastrointestinal Symptom score; Visual Analogue Scale; Functional Dyspepsia-related Quality of Life; Electrogastrography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Banhasasim-tang (Experimental)
  Interventions: Dietary Supplement: Banhasasim-tang
- Placebo drug (Placebo Comparator): The placebo of this study is corn-starch granules. It has the same form, color, flavor and amount like experimental herbal extracted formula
  Interventions: Dietary Supplement: Corn-starch granules

INTERVENTIONS:
Dietary Supplement: Banhasasim-tang — Form : granules Contents : It consists of seven Herbs. It contains Rhizoma Pinelliae, Radix Scutellariae, Zingiberis Rhizoma, Panax ginseng, Glycyrrhiza uralensis Fisch, Zizyphi Fructus and Coptidis Rhizoma Dosage and frequency : 9g per day (three times a day) Route of administration : Oral Administration duration : 42 days in the study
  Other Names: Brand names : Bansasin granules
  Arms: Banhasasim-tang
Dietary Supplement: Corn-starch granules — This placebo has the same form, color, and flavor as experimental intervention.The dosage, frequency and duration is also same as experimental intervention.
  Other Names: Corn-starch granules with herb decoctions flavor
  Arms: Placebo drug

SUMMARY:
The purpose of this study is to assess efficacy based on Gastrointestinal Symptom score and safety based on the rate of adverse event or laboratory findings of Banhasasim-tang administrated three times a day orally on functional dyspepsia.

DETAILED DESCRIPTION:
Banhasasim-tang

1. Main 3 gram herb powder (including Rhizoma Pinelliae, Radix Scutellariae, Zingiberis Rhizoma, Panax ginseng, Glycyrrhiza uralensis Fisch, Zizyphi Fructus and Coptidis Rhizoma) of old oriental prescriptions for dyspepsia.
2. Usually having used for dyspepsia in asia
3. Need for correct clinical information by RCT

ELIGIBILITY:
Inclusion Criteria:

1. Typical functional dyspepsia according to ROME III criteria.

   * One or more of:

     * Bothersome post-prandial fullness
     * Early satiation
     * Epigastric pain
     * Epigastric burning
   * No evidence of structural disease (including at upper endoscopy) that is likely to explain the symptoms
2. The presence of 'moderate' as the degree of severity for at least three Gastrointestinal Symptom (GIS) score symptoms
3. Before participation of trial, epigastric pain or discomfort has persisted in a permanent or recurrent form for a minimum period of 12 weeks
4. Written and informed consent

Exclusion Criteria:

1. History of peptic ulcer or gastroesophageal reflux disease(GERD)
2. Current prominent symptoms of irritable bowel syndrome or GERD
3. Presence of the following alarm symptoms:

   * Severe weight loss
   * Black or tar stool
   * Dysphagia
4. Presence of the following diseases (like cholangitis, pancreatitis, etc.) or uncontrolled severe organ disorders
5. Women in pregnancy and lactation
6. History of gastrointestinal surgery or taking any drugs that may significantly alter digestive system
7. Participation of other clinical trials within the last 3 months
8. Severe mental problems or drug abuse
9. Judged by expert that they are appropriate to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom (GIS) score (epigastric pain/upper abdominal pain, abdominal cramps, fullness, early satiety, loss of appetite, sickness, nausea, vomiting, retrosternal discomfort, and acidic regurgitation/heartburn) | Baseline, 2 weeks, 4 weeks, 6 weeks after administration, 4 and 8 weeks after treatment finish

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) for overall discomfort due to dyspepsia | Baseline, 2weeks, 4weeks, 6weeks after administration, 4 and 8 weeks after treatment finish
Functional Dyspepsia-related Quality of Life (FD-QoL) | Baseline, 2 weeks, 4 weeks, and 6 weeks after administration, 4 and 8 weeks after treatment finish
Electrogastrography (EGG) | Baseline, 6 weeks after administration

CONTACTS AND LOCATIONS:
Overall Officials: Jin-sung Kim, Ph.D, Principal Investigator — Kyung Hee University Medical Center Oriental Hospital
Locations (2):
- South Korea (2):
  - Kyung Hee University Medical Center Oriental Hospital, Seoul
  - East-West Neo Medical Center, Seoul

REFERENCES:
- [Derived] Park JW, Ryu B, Yeo I, Jerng UM, Han G, Oh S, Lee J, Kim J. Banha-sasim-tang as an herbal formula for the treatment of functional dyspepsia: a randomized, double-blind, placebo-controlled, two-center trial. Trials. 2010 Jul 30;11:83. doi: 10.1186/1745-6215-11-83. PMID 20670451